CLINICAL TRIAL: NCT07171229
Title: Evaluation of Cytokines Level as an Indicator of Pulp Inflammation and Its Relation to the Success Rates of Pulpotomy in Primary Molars Affected With Proximal Versus Occlusal Decay: Non-Randomized Clinical Trial
Brief Title: Evaluation of Cytokines Level as an Indicator of Pulp Inflammation and Its Relation to the Success Rates of Pulpotomy in Primary Molars Affected With Proximal Versus Occlusal Decay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Khalifa, PHD candidate, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14422023529314
Record Dates: First submitted 2025-08-25; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pulpitis - Reversible; Occlusal Caries; Proximal Caries
Keywords: pulpotomy; cytokines
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusal decay (Experimental): Primary molars diagnosed with reversible pulpits caused by occlusal decay
  Interventions: Procedure: Pulpotomy; Other: Measuring Cytokines level
- Proximal decay (Active Comparator): Primary molars diagnosed with reversible pulpits caused by Proximal decay.
  Interventions: Procedure: Pulpotomy; Other: Measuring Cytokines level

INTERVENTIONS:
Procedure: Pulpotomy — * Local anesthesia will be administered, and the tooth will be isolated with a rubber dam.
  * To minimize further bacterial contamination, carious tissues will be removed progressively, starting from the cavity periphery and then over the pulp chamber roof.
  * Before managing the pulpal hemorrhage, a sterile cotton pellet will be placed over the pulp tissue for 30-45 s.
  * A fresh sterile bur will be used to remove all coronal pulp tissue down to the root canal orifices, with copious water irrigation
  * MTA will be used as medicament of choice for pulpotomy.
  * The pulpotomy-treated tooth will be prepared to receive a full-coverage stainless steel crown (SSC) after the procedure.
Other: Measuring Cytokines level — measuring cytokines level as an indicator for pulp inflammation

SUMMARY:
pulpotomy will be done I primary molars with occlusal or proximal decay and level of cytokines will be measured as an indicator for pulp inflammation levels

DETAILED DESCRIPTION:
The proposed trial interventions, pulpotomy, will follow standard clinical procedural guidelines. Participants will be allocated to one of the two intervention groups only after intra-operative confirmation of pulp vitality and achievement of radicular pulp hemostasis.

Standard clinical protocol for both groups with occlusal and proximal decay:

1. A detailed history of symptoms will be obtained, and a thorough clinical examination will be conducted.
2. Pre-operative pain intensity will be assessed using a validated five-face visual analog scale (VAS), where children select the face that best represents their pain level.
3. A standard pre-operative periapical radiograph will be taken, ensuring the image extends beyond the root tip and shows no distortion or processing errors.
4. Local anesthesia will be administered, and the tooth will be isolated with a rubber dam.
5. To minimize further bacterial contamination, carious tissues will be removed progressively, starting from the cavity periphery and then over the pulp chamber roof.
6. Before managing the pulpal hemorrhage, a sterile cotton pellet will be placed over the pulp tissue for 30-45 s. to obtain pulpal blood samples. The specimens will be collected into heparin-coated tubes with 1 mg saline solution and stored at - 20 °C (-4.0 °F) for 6 months until the day of testing.
7. A fresh sterile bur will be used to remove all coronal pulp tissue down to the root canal orifices, with copious water irrigation. Intra-operative assessment of pulp vitality will be conducted, with healthy vital pulp appearing as uniformly reddish-pink vascular tissue and non-vital pulp as dark avascular tissue or yellowish liquefied areas. If necrotic, the tooth will be excluded from the study, and local management protocols will be followed for treatment (Bas et al., 2024).
8. MTA will be used as medicament of choice for pulpotomy.
9. Once a 2-3 mm thickness is ensured, the cavity will be filled with restorative glass ionomer cement to seal it.
10. The pulpotomy-treated tooth will be prepared to receive a full-coverage stainless steel crown (SSC) after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children with provoked pain.
* Caries in proximal surface to the dentine full thickness.
* Caries in occlusal surface to the dentine full thickness.
* Radicular pulp health is verified by achieving hemostasis within eight minutes of compression using a cotton pellet with 5% sodium hypochlorite.

Exclusion Criteria:

* Unrestorable primary molars.
* Primary molars with spontaneous pain.
* Medically compromised patients who have systemic disease.
* Uncooperative children who refuse treatment.
* Children whose parents are unwilling to place stainless steel crowns.
* Children whose parents or caregivers refuse to participate in the study or are unable to attend follow-up visits.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Post operative Pain | pain will be measured at one week , 3 months , 6 months and 12 months.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).
Preapical lesion | will be measured at 3 months , 6 months and 12 months
  by Clinical examination: presence of Swelling, sinus tract, or fistula: ,(binary outcome: present or absent )
Pain on percussion | will be measured at 3 months , 6 months and 12 months
  Tapping the tooth with the blunt end of the mirror binary outcome: present or absent
Mobility | will be measured at 3 months , 6 months and 12 months
  using Miller's mobility test :involves holding the tooth firmly between two instruments and assessing its mobility on a scale from 0 to 3. A score of 0 indicates no detectable movement, while scores of 1-3 represent increasing degrees of mobility.
  it will be measured as present for any score from 1 to 3 (binary: present or absent)

SECONDARY OUTCOMES:
radiographic success | baseline data at the first visit following the procedure completion and at 6 and 12 months
  using Digital periapical intraoral radiograph
  Radiographic Success:
  • Radiolucency at the furcation or periapical area, internal or external root resorption, will be examined (present or not) through digital periapical radiographs.
  Criteria for radiographic success
  * No evidence of extensive pathologic root resorption.
  * No evidence of pathological interradicular and/or periapical radiolucency.
  * No evidence of the development of pathologic radiolucency involving the successor tooth germ.
Cytokines level | at the time of pulpotomy procedure
  blood sample will be collected from exposed pulp chamber before removal and IL-8 & IL-10 levels will be measured using Enzyme-linked immunoassay ( ELISA) kit. unit of measurement: ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Hany Saber, Study Chair — Professor of Pediatric Dentistry, Faculty of dentistry, Cairo Univeristy; Maii Mohammed, Study Director — lecturer of Pediatric Dentistry, Faculty of dentistry, Cairo Univeristy; Yasmin Magdi Khalifa, Principal Investigator
Locations (1):
- Cairo Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No